CLINICAL TRIAL: NCT03924076
Title: Effect of Paraprobiotic Lactobacillus Plantarum IS-10506 on Humoral Immune Response of Indonesian Elementary School Children: a Double Blind, Randomized, Placebo-controlled Trial
Brief Title: Effect of Paraprobiotic Lactobacillus Plantarum IS-10506 on Humoral Immune Response of Elementary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, DR.Siti Helmyati, DCN, M.Kes, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KE/FK/293/EC/2018
Record Dates: First submitted 2019-04-16; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Humoral Immune Response

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Received UHT milk + paraprobiotic Lactobacillus plantarum IS-10506 5 x 1010 CFU/day (125 mL) for 90 days
  Interventions: Dietary Supplement: UHT Milk + Lactobacillus plantarum IS-10506
- Placebo Group (Placebo Comparator): Received UHT milk (125 mL) for 90 days
  Interventions: Dietary Supplement: UHT Milk

INTERVENTIONS:
Dietary Supplement: UHT Milk + Lactobacillus plantarum IS-10506 — 125 ml UHT milk (+Lactobacillus plantarum IS-10506) given to treatment group
  Arms: Treatment Group
Dietary Supplement: UHT Milk — 125 ml UHT milk given to placebo group
  Arms: Placebo Group

SUMMARY:
This study is aimed to determine effect of paraprobiotic Lactobacillus plantarum IS-10506 on humoral immune response by measuring faecal sIgA and blood IgG, IgM, and IgA

DETAILED DESCRIPTION:
The type of the study is double blind randomize placebo-controlled trial with minimum 72 subjects which divided into 2 groups i.e. 1) placebo group which will receive UHT milk (125 mL) and 2) treatment group which will received UHT milk + paraprobiotic Lactobacillus plantarum IS-10506 5 x 1010 CFU/day (125 mL). The subjects have to consume one pack of milk every day for 90 consecutive days. Before and after intervention (day 30 and day 90), several data will be collected i.e. faecal sIgA, blood IgG, IgM, and IgA. The subjects recruited from elementary school in Yogyakarta District.

ELIGIBILITY:
Inclusion Criteria:

* children at age of 7-9 years
* have normal body mass index (BMI) i.e. -2 ≤ z-score < +1, slightly overweight z-score < +1.5, and slightly underweight z-score > -3.

Exclusion Criteria:

* allergic to milk
* consuming other probiotic product
* he/she do not want to stop consumption & doing washout for 2 weeks.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Serum IgG | 90 days
  Measuring IgG (ng/mL) in collected serum
Serum IgA | 90 days
  Measuring IgA (ng/mL) in collected serum
Serum IgM | 90 days
  Measuring IgM (ng/mL) in collected serum
Faecal sIgA | 90 days
  Measuring sIgA (ng/mL) in collected feses

SECONDARY OUTCOMES:
Weight | 90 days
  Measuring weight (kg) change
Height | 90 days
  Measuring height (cm) change

CONTACTS AND LOCATIONS:
Overall Officials: Siti Helmyati, DR., Principal Investigator — Gadjah Mada University; Mohammad Juffrie, Prof.dr., Principal Investigator — Gadjah Mada University; Lily A Lestari, DR., Principal Investigator — Gadjah Mada University
Locations (1):
- Universitas Gadjah Mada, Sleman, D.I.Yogyakarta, Indonesia